CLINICAL TRIAL: NCT06631378
Title: The Incidence of Surgical Site Complications in Transverse Versus Longitudinal Groin Incision in Vascular Surgery: A Randomized Clinical Trial
Brief Title: Transverse Versus Longitudinal Groin Incision in Vascular Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kolding Sygehus (Other)
Collaborators: Region of Southern Denmark (Other); University of Southern Denmark (Other)
Responsible Party: Principal Investigator, Christina Pilgaard Madsen, MD, PhD-student, Kolding Sygehus
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KoldingSygehusKarkir
Record Dates: First submitted 2024-09-27; First posted 2024-10-08 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-03

CONDITIONS: Peripheral Arterial Disease(PAD); Aneurysmal Disease
Keywords: groin wound complications; surgical site complications; surgical site complication; vascular surgery; incision type; incision
MeSH Terms: conditions — Peripheral Arterial Disease; Surgical Wound

STUDY DESIGN:
Intervention Model Description: The trial is a single center superiority randomized clinical trial with two parallel groups with 1:1 randomization to either transverse or longitudinal incision in the groin in vascular surgery with arterial reconstruction.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transverse groin incision (Experimental)
  Interventions: Procedure: Transverse groin incision
- Longitudinal groin incision (Active Comparator)
  Interventions: Procedure: Longitudinal incision

INTERVENTIONS:
Procedure: Transverse groin incision — The transverse incision is made parallel to the inguinal ligament either superiorly or inferiorly to the skin crease directly over the femoral artery. The subcutaneous tissue is dissected in the transverse direction till Scarpaes fascia after which the dissection is performed in the longitudinal direction along the line of the vessels. The lymphatic vessels are spared as much as possible. Any damaged lymph vessels are closed with surgical clips. Damages lymph nodes are either removed or the capsule is sutured to prevent lymph leakage. In case of difficulty with proper access to the femoral arteries, the incision can be extended either medially, laterally, or vertically.
  Arms: Transverse groin incision
Procedure: Longitudinal incision — The longitudinal incision is made directly over the femoral artery from the inguinal ligament. The subcutaneous tissue is dissected along the line of the vessel sparing the lymphatic vessels as much as possible. Any damaged lymph vessels are closed with clips. Damages lymph nodes are either removed or the capsule is sutured to prevent lymph leakage.
  Arms: Longitudinal groin incision

SUMMARY:
The purpose of the study is to examine whether incision type has an influence on the development of groin wound complications after operation in the groin in vascular surgery.

The main questions it aims to answer are:

Does a transverse incision in the groin lead to fewer surgical site complications than a longitudinal incision? Does a transverse incision lead to fewer readmissions, fewer reoperations, shorter length of hospital stay, and a lower amputation rate.

Participants will undergo vascular surgery in the groin with either a transverse or longitudinal incision. The incision type will be selected randomly.

ELIGIBILITY:
Inclusion Criteria:

• Patients undergoing vascular reconstruction with a groin incision

Exclusion Criteria:

* Patients previously operated with a groin incision.
* Patients undergoing operation due to trauma, bleeding, or pseudoaneurysm.
* Patients operated within the first 24 hours of admission.
* If it prior to the operation is deemed necessary with a muscleplasty.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 232 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of surgical site complications | 35 days after the operation
  The surgical site complications are defined as follows:
  * Surgical site infection according to the Szilagy classification:
  * Dehiscence with separation of the wound edges and exposure of the underlying tissue.
  * Lymhocele defined as the presence of localized swelling in the groin and verified on ultrasound as an anechoic fluid collection.
  * Hematoma defined as the presence of localized swelling in the groin with discoloration and verified on ultrasound as an echoic fluid collection.

SECONDARY OUTCOMES:
Reoperation | 35 days after the operation
  Reoperation in the groin due to surgical site complications Reoperation due to the reconstruction Minor or major amputation
Readmission | 35 days
  Is the patient readmitted due to either surgical site complications or for other reasons
• Length of stay | 35 days
  The duration of the hospital stay after the operation.
Mortality | 35 days
  Death and the cause of death.
Healing of the groin | 35 days
  Evaluation of the groin to access if it has healed irrespective of the development of surgical site complications.

CONTACTS AND LOCATIONS:
Overall Officials: Kim Trine Maria Mejnert Jørgensen, MD, PhD, Study Director — Department of vascular surgery, Kolding Hospital
Locations (1):
- Department of Vascular Surgery - Lillebaelt Hospital, Kolding, Denmark

IPD SHARING:
Plan to Share IPD: No